CLINICAL TRIAL: NCT02326363
Title: Mindfulness-Based Recovery in Veterans With Substance Use Disorders
Brief Title: Mindfulness-Based Recovery in Veterans
Acronym: MBR-Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D1292-R; I01RX001292 (NIH)
Record Dates: First submitted 2014-12-22; First posted 2014-12-29 (Estimated); Results first posted 2020-07-10 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-01

CONDITIONS: Substance Abuse; Depression; Anxiety Disorder
Keywords: substance abuse; Mental Health Disorders
MeSH Terms: conditions — Substance-Related Disorders; Depression; Anxiety Disorders

STUDY DESIGN:
Masking Description: No masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mindfulness Based Relapse Prevention (MBRP): (Experimental): The Introductory session provides an orientation to the intervention, basic mindfulness techniques and general description of group sessions. Each session has a central theme/topic and consists of in-session experiential practice, discussions and homework assignments. Sessions begin with a check-in followed by a 20-30 minute meditation (i.e. body scan). The therapist reviews homework assignments, discusses challenges and participants are taught a variety of mindfulness meditation (MM) practices such as breath meditation, urge surfing, walking or movement meditation.
  Interventions: Behavioral: Mindfulness Based Relapse Prevention (MBRP)
- Twelve-Step Facilitation Intervention (TSF) (Active Comparator): The Introductory session covers the 12-Step view of addiction and therapy overview. The manual, originally developed for individual sessions, has been adapted for group delivery. The eight selected sessions include four topics chosen by the manual developers as core topics and four elective topics. The intervention involves helping participants understand and incorporate core principles of 12-Step approaches while encouraging active participation in 12-Step meetings and related activities. The primary goal is to promote abstinence by facilitating the patient's acceptance and surrender of addiction. Sessions begin with a check-in during which participants introduce themselves, report on meeting attendance and participation in related activities, any alcohol/drug use or craving to use. The remainder of the session focuses on discussion of the topic content followed by a "take home" summary and homework assignment.
  Interventions: Behavioral: Twelve-Step Facilitation Intervention (TSF)

INTERVENTIONS:
Behavioral: Mindfulness Based Relapse Prevention (MBRP) — Each session has a central theme/topic and consists of in-session experiential practice, discussions and homework assignments. Sessions begin with a check-in followed by a 20-30 minute meditation (i.e. body scan). The therapist reviews homework assignments, discusses challenges and participants are taught a variety of MM practices such as breath meditation, urge surfing, walking or movement meditation.
  Arms: Mindfulness Based Relapse Prevention (MBRP):
Behavioral: Twelve-Step Facilitation Intervention (TSF) — The primary goal is to promote abstinence by facilitating the patient's acceptance and surrender of addiction. Sessions begin with a check-in during which participants introduce themselves, report on meeting attendance and participation in related activities, any alcohol/drug use or craving to use. The remainder of the session focuses on discussion of the topic content followed by a "take home" summary and homework assignment.
  Arms: Twelve-Step Facilitation Intervention (TSF)

SUMMARY:
This study will provide important information concerning the used of mindfulness-based relapse prevention (MBRP) as a continuing care strategy for Veterans who have completed primary treatment for a SUD. Most research is focused on the acute care of SUDs, but the risk of relapse to substance use is highest during the period immediately following treatment and attention to continuing care is critical. If this trial demonstrates that MBRP promotes sustained abstinence and improved functional outcomes, this will provide a valuable treatment to facilitate rehabilitation and recovery for Veterans with SUDs.

DETAILED DESCRIPTION:
Rates of substance use disorders (SUDS) are high among military personnel and Veterans. While much research is focused on the acute care of SUDs, the risk of relapse to substance use following treatment is high and attention to continuing care is critical. New continuing care strategies targeting life-style change and improved coping mechanisms are important in facilitating maintenance of abstinence, promoting rehabilitation and functional recovery for Veterans with SUDs. Mindfulness-based relapse prevention (MBRP), a manualized treatment integrating cognitive-behavioral relapse prevention therapy with mindfulness practices, has shown promise in continuing care for SUDs. The proposed project will compare MBRP to a 12-Step Facilitation treatment as a continuing care strategy following primary treatment for SUDs. Participants will be randomized to participate in 8-weeks of weekly 90-minute, group-based MBRP or 12-Step Facilitation followed by a 10-month follow-up period with regular assessments of substance use, mood/anxiety symptoms, quality of life and functional outcomes. Two VAMC sites (Charleston and Tuscaloosa) with a history of successful collaboration will work together to recruit an adequate sample size to address the primary study questions within a 4-year period and to ensure generalizability of the results. If this trial demonstrates that MBRP promotes sustained abstinence and improved functional outcomes, this will provide a valuable treatment to facilitate rehabilitation and recovery for Veterans with SUDs.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women military Veterans who have completed the Charleston or Tuscaloosa Veterans Administration Medical Center (VAMC) intensive outpatient substance abuse treatment program, a residential treatment program, or an intensive outpatient program similar to the Charleston or Tuscaloosa VAMC program.
2. Able to comprehend English.
3. Meets DSM-V criteria for a current substance use disorder and have used substances in the 30 days prior to treatment entry. Participants on medications targeting their substance use must be stabilized on medications for at least 2 weeks before therapy initiation.
4. May meet criteria for a mood, anxiety or other psychiatric disorder. Participants on maintenance medications for a mood or anxiety disorder must be stabilized on medications for at least 2 weeks before therapy initiation.
5. Able to adequately provide informed consent and function at an intellectual level sufficient to allow accurate completion of all assessment instruments.
6. Willing to commit to 8 group therapy sessions, baseline, weekly and follow-up assessments for 10-months after the end of treatment (12-month total).

Exclusion Criteria:

1. Active suicidal or homicidal ideation with a plan as this is likely to require hospitalization or other interventions that could interfere with study participation.
2. Unstable psychiatric condition likely to require hospitalization or other interventions that would interfere with study participation.
3. Unstable medical condition or one that may require hospitalization during the course of the study.
4. Meets criteria for nicotine dependence only
5. Women who are pregnant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2015-03-16 (Actual); Primary Completion 2018-10-29 (Actual); Study Completion 2018-10-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Theresa Brady, MD PhD, Principal Investigator — Ralph H. Johnson VA Medical Center, Charleston, SC
Locations (2):
- United States (2):
  - Tuscaloosa VA Medical Center, Tuscaloosa, AL, Tuscaloosa, Alabama
  - Ralph H. Johnson VA Medical Center, Charleston, SC, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Killeen TK, Baker NL, Davis LL, Bowen S, Brady KT. Efficacy of mindfulness-based relapse prevention in a sample of veterans in a substance use disorder aftercare program: A randomized controlled trial. J Subst Use Addict Treat. 2023 Sep;152:209116. doi: 10.1016/j.josat.2023.209116. Epub 2023 Jun 25. PMID 37364669
- [Derived] Brady KT, Killeen T, Baker NL. Efficacy of mindfulness-based relapse prevention in veterans with substance use disorders: Design and methodology of a randomized clinical trial. Contemp Clin Trials. 2021 Jun;105:106393. doi: 10.1016/j.cct.2021.106393. Epub 2021 Apr 20. PMID 33857680

RESULTS

PARTICIPANT FLOW:
Groups:
- Mindfulness Based Relapse Prevention (MBRP):: Mindfulness Based Relapse Prevention (MBRP): Each session has a central theme/topic and consists of in-session experiential practice, discussions and homework assignments. Sessions begin with a check-in followed by a 20-30 minute meditation (i.e. body scan).
- Twelve-Step Facilitation Intervention (TSF): The Introductory session covers the 12-Step view of addiction and therapy overview. The manual, originally developed for individual sessions, has been adapted for group delivery (Brown et al., 2002). The eight selected sessions include four topics chosen by the manual developers as core topics and four elective topics.
Period: Overall Study
Arm/Group | Mindfulness Based Relapse Prevention (MBRP): | Twelve-Step Facilitation Intervention (TSF)
Started | 98 | 106
Completed | 47 | 50
Not Completed | 51 | 56

BASELINE CHARACTERISTICS:
Population: 237 consented and screened individuals, 204 were randomized (n=98 to MM and n=106 to TAU)
Groups:
- Total: Total of all reporting groups
Arm/Group | Mindfulness Based Relapse Prevention (MBRP): | Twelve-Step Facilitation Intervention (TSF) | Total
Number analyzed (Participants) | 98 | 106 | 204
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.1 (9.8) | 54.2 (10) | 53.2 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 92 | 100 | 192
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 78 | 86 | 164
  White | 15 | 15 | 30
  More than one race | 3 | 1 | 4
  Unknown or Not Reported | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  United States | 98 | 106 | 204
Study Site [Count of Participants; unit: Participants]
  Charleston SC VA | 58 | 62 | 120
  Birmingham AL VA | 40 | 44 | 84

OUTCOME MEASURES:

1. Primary Outcome: Timeline Follow-Back (TLFB) - Number of Participants With Alcohol, Illicit Substance and Cigarette Use During Treatment up to 8 Weeks. Available Date
Description: The TLFB will be used to obtain retrospective self-report of alcohol and illicit drug (e.g., cocaine, marijuana, stimulants, sedatives, opioids) use using calendar and memory prompts to stimulate recall. The TLFB yields consistently high test-retest correlations and correlates well with other self-reports and collateral reports. Quantity and frequency assessments as well as time-to-event measures can be obtained. Drug/alcohol use in treatment up to 8 weeks will be assessed.
Time Frame: Study Treatment Duration up to 8 Weeks
Population: participants randomized and reporting use/no with at least 1 treatment visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Mindfulness Based Relapse Prevention (MBRP): | Twelve-Step Facilitation Intervention (TSF)
Number analyzed (Participants) | 74 | 87
Participants
  Any Alcohol Use During Study Treatment | 8 | 12
  Any Illicit Substance Use During Study Treatment | 9 | 4
  Cigarette Use During Study Treatment | 46 | 62

2. Primary Outcome: Timeline Follow-Back (TLFB) - Number of Participants With Alcohol, Binge Alcohol, Illicit Drug Use. Available Date
Description: The TLFB will be used to obtain retrospective self-report of alcohol and illicit drug (e.g., cocaine, marijuana, stimulants, sedatives, opioids) use using calendar and memory prompts to stimulate recall. The TLFB yields consistently high test-retest correlations and correlates well with other self-reports and collateral reports (Carey, 1997). Quantity and frequency assessments as well as time-to-event measures can be obtained. Drug/alcohol use during treatment through10 months will be assessed.
Time Frame: Study Treatment Duration through 10 Months Follow up
Population: Any alcohol, binge alcohol or illicit substance use reported during study treatment through 10 months.
  Available Data
Measure: Count of Participants; unit: Participants
Arm/Group | Mindfulness Based Relapse Prevention (MBRP): | Twelve-Step Facilitation Intervention (TSF)
Number analyzed (Participants) | 98 | 106
Participants
  Any Alcohol Use | 25 | 37
  Any Binge Alcohol Use | 13 | 20
  Any Illicit Substance Use | 18 | 29

3. Primary Outcome: Time to Relapse to Substance Use - Days to First Alcohol, Binge Alcohol and Illicit Substance Use. Available Data
Description: The TLFB will be used to obtain retrospective self-report of alcohol and illicit drug (e.g., cocaine, marijuana, stimulants, sedatives, opioids) use using calendar and memory prompts to stimulate recall. The TLFB yields consistently high test-retest correlations and correlates well with other self-reports and collateral reports. Quantity and frequency assessments as well as time-to-event measures can be obtained. Participants that failed to return for any treatment or follow up visits are considered censored at study day 1.
Time Frame: Study Treatment Duration through 10 Months
Measure: Median (Inter-Quartile Range); unit: Days to first relapse
Arm/Group | Mindfulness Based Relapse Prevention (MBRP): | Twelve-Step Facilitation Intervention (TSF)
Number analyzed (Participants) | 98 | 106
Days to first relapse
  Relapse to any Alcohol Use | 110 [74 to 138] | 128 [45 to 195]
  Relapse to Binge Alcohol Use | 95 [78 to 135] | 196 [94 to 298]
  Relapse to any Illicit Substance Use | 1 [1 to 265] | 48 [1 to 293]

4. Secondary Outcome: Mindfulness Acceptance and Awareness Scale (MAAS)
Description: This is a 15-item self-report instrument rating the frequency of experiencing impaired moment-to-moment attention on a 6-point Likert scale. Scores range from 1- 6 with higher scores indicating higher levels of mindfulness. This measure explores the relationship between MAAS scores and treatment response.
Time Frame: Baseline, End of treatment, 3 Months, 6 Months, 10 Months
Population: data are reported as those available at study baseline and each subsequent study outcome time point.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Mindfulness Based Relapse Prevention (MBRP): | Twelve-Step Facilitation Intervention (TSF)
Number analyzed (Participants) | 98 | 106
units on a scale
  Baseline | 3.99 (0.10) | 4.12 (0.1)
  End of Treatment: number analyzed (Participants) | 51 | 66
  End of Treatment | 4.04 (0.12) | 4.26 (0.14)
  3 Months: number analyzed (Participants) | 49 | 55
  3 Months | 4.10 (0.14) | 4.55 (0.15)
  6 Months: number analyzed (Participants) | 46 | 50
  6 Months | 3.93 (0.17) | 4.49 (0.16)
  10 Months: number analyzed (Participants) | 46 | 48
  10 Months | 4.02 (0.17) | 4.58 (0.17)

5. Secondary Outcome: Beck Depression Inventory 2
Description: This 21-item self-report scale will be used to assess for worsening depression/suicidality in safety monitoring. Scores range from 0 - 63 with higher scores indicating more severe depression.
Time Frame: Baseline, End of Treatment, 3 Months, 6 Months, 10 Months
Population: data are reported as those available at study baseline and each subsequent study outcome time point.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Mindfulness Based Relapse Prevention (MBRP): | Twelve-Step Facilitation Intervention (TSF)
Number analyzed (Participants) | 98 | 106
units on a scale
  Baseline | 15.28 (0.97) | 14.26 (0.95)
  End of Treatment: number analyzed (Participants) | 50 | 66
  End of Treatment | 8.96 (1.12) | 7.02 (0.97)
  3 Months: number analyzed (Participants) | 48 | 54
  3 Months | 11.75 (1.28) | 8.93 (1.24)
  6 Months: number analyzed (Participants) | 46 | 50
  6 Months | 12.02 (1.28) | 9.50 (1.29)
  10 Months: number analyzed (Participants) | 46 | 48
  10 Months | 12.15 (1.44) | 9.17 (1.33)

6. Secondary Outcome: Beck Anxiety Inventory
Description: This 21-item self-report scale has symptom clusters reflecting neurophysiological, subjective, panic, and autonomic dimensions. Scores range from 0-63 with higher scores indicating more severe anxiety.
Time Frame: Baseline, End of Treatment, 3 Months, 6 Months, 10 Months
Population: data are reported as those available at study baseline and each subsequent study outcome time point.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Mindfulness Based Relapse Prevention (MBRP): | Twelve-Step Facilitation Intervention (TSF)
Number analyzed (Participants) | 98 | 106
units on a scale
  Baseline | 14.99 (1.22) | 16.28 (1.42)
  End of Treatment: number analyzed (Participants) | 49 | 106
  End of Treatment | 14.94 (1.64) | 11.09 (1.65)
  3 Months: number analyzed (Participants) | 49 | 106
  3 Months | 14.24 (1.74) | 10.46 (1.8)
  6 Months: number analyzed (Participants) | 44 | 106
  6 Months | 14.2 (1.76) | 11.40 (1.53)
  10 months: number analyzed (Participants) | 46 | 106
  10 months | 14.15 (1.72) | 12.90 (1.91)

7. Secondary Outcome: Urine Drug Screen
Description: Observed urine samples will be collected with a RapidCHECK Multi-Drug 10 Panel Test, which allows detection of tetrahydrocannabinol (THC)/marijuana, cocaine, phencyclidine, opiates, methamphetamines, methadone, amphetamines, barbiturates, benzodiazepines and uses concentrations levels established by the National Institute on Drug Abuse (NIDA) and the World Health Organization (WHO). Osmolality and temperature assessed at collection time to insure sample validity.
Time Frame: Weekly, Week 8, 3 Months, 6 Months, 10 Months
Population: Intent to Treat Sample of those with positive urine drug screens for THC
Measure: Count of Participants; unit: Participants
Arm/Group | Mindfulness Based Relapse Prevention (MBRP): | Twelve-Step Facilitation Intervention (TSF)
Number analyzed (Participants) | 98 | 106
Participants
  Week 1: number analyzed (Participants) | 67 | 93
  Week 1 | 0 | 0
  Week 2: number analyzed (Participants) | 67 | 76
  Week 2 | 1 | 3
  Week 3: number analyzed (Participants) | 59 | 75
  Week 3 | 2 | 2
  Week 4: number analyzed (Participants) | 51 | 68
  Week 4 | 0 | 2
  Week 5: number analyzed (Participants) | 54 | 65
  Week 5 | 0 | 1
  Week 6: number analyzed (Participants) | 48 | 61
  Week 6 | 0 | 1
  Week 7: number analyzed (Participants) | 37 | 60
  Week 7 | 0 | 2
  Week 8: number analyzed (Participants) | 49 | 64
  Week 8 | 0 | 3
  3 Months: number analyzed (Participants) | 50 | 53
  3 Months | 3 | 5
  6 Months: number analyzed (Participants) | 43 | 45
  6 Months | 2 | 6
  10 Months: number analyzed (Participants) | 44 | 49
  10 Months | 8 | 6

8. Secondary Outcome: EtG
Description: The conjugated alcohol metabolite ethyl glucuronide (EtG) remains positive in urine for several days following cessation and is a useful biomarker of recent drinking in outpatient settings (Dahl 2011). This will be used as the primary biologic assessment of drinking status as breathalyzer tests only assess very recent alcohol use. The assay will be done in the Charleston VAMC laboratory on samples collected at baseline, end of treatment and 3-, 6-, and 10-month follow-up visits.
Time Frame: Week 8, 3 Months, 6 Months, 10 Months
Population: Data listed as those with a positive EtG reading at each visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Mindfulness Based Relapse Prevention (MBRP): | Twelve-Step Facilitation Intervention (TSF)
Number analyzed (Participants) | 98 | 106
Participants
  Week 8: number analyzed (Participants) | 49 | 63
  Week 8 | 4 | 9
  3 Month: number analyzed (Participants) | 50 | 53
  3 Month | 3 | 1
  6 Month: number analyzed (Participants) | 43 | 45
  6 Month | 2 | 1
  10 Month: number analyzed (Participants) | 44 | 49
  10 Month | 1 | 1

9. Secondary Outcome: Addiction Severity Index, Lite
Description: This standardized, multidimensional, semi-structured interview provides information concerning functioning in six domains commonly impacted by substance abuse: alcohol/drug, medical, psychiatric, legal, family/social and employment. The alcohol/drug scale composite score will be reported to determine severity of alcohol/drug problem severity. The average range is 0 (denoting a better outcome) to 1 ( denoting a worse outcome).
Time Frame: 8 Weeks, 3 Months, 6 Months, 10 Months
Population: some participants missed certain follow-ups.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Mindfulness Based Relapse Prevention (MBRP): | Twelve-Step Facilitation Intervention (TSF)
Number analyzed (Participants) | 52 | 65
score on a scale
  8 Weeks: number analyzed (Participants) | 50 | 65
  8 Weeks | .1186 (.1209) | .1180 (.1368)
  3 Months: number analyzed (Participants) | 51 | 55
  3 Months | .1115 (.1651) | .0877 (.1452)
  6 Months: number analyzed (Participants) | 48 | 52
  6 Months | .0764 (.1502) | .1124 (.1721)
  10 Months: number analyzed (Participants) | 52 | 53
  10 Months | .0806 (.1215) | .1212 (.1428)

10. Secondary Outcome: Days Engaging in Structured/Productive Work Activities (PWAC)
Description: The PWAC will be used to assess self-reported days engaged in structured, volunteer, or employed work activity of at least 1 hour in duration. VISTA queries using Compensated Work Therapy and Veterans Enrichment Program stop codes will be run for medical record corroboration. Activities outside of the VA will be included.
Time Frame: Weekly, Week 8, 3 Months, 6 Months, 10 Months
Population: data are reported as those available at each study outcome time point.
Measure: Median (Inter-Quartile Range); unit: days reported
Arm/Group | Mindfulness Based Relapse Prevention (MBRP): | Twelve-Step Facilitation Intervention (TSF)
Number analyzed (Participants) | 98 | 106
days reported
  Week 1: number analyzed (Participants) | 98 | 93
  Week 1 | 1 [0 to 4] | 0 [0 to 3]
  Week 2: number analyzed (Participants) | 98 | 78
  Week 2 | 0 [0 to 5] | 0 [0 to 3]
  Week 3: number analyzed (Participants) | 98 | 77
  Week 3 | 2 [0 to 6] | 0 [0 to 3]
  Week 4: number analyzed (Participants) | 98 | 68
  Week 4 | 2 [0 to 6] | 1 [0 to 5]
  Week 5: number analyzed (Participants) | 98 | 66
  Week 5 | 2 [0 to 7] | 1 [0 to 5]
  Week 6: number analyzed (Participants) | 98 | 62
  Week 6 | 3 [0 to 6] | 1 [0 to 5]
  Week 7: number analyzed (Participants) | 98 | 61
  Week 7 | 2 [0 to 6] | 1 [0 to 5]
  Week 8: number analyzed (Participants) | 98 | 68
  Week 8 | 2.5 [0 to 7] | 1 [0 to 7.5]
  3 Months: number analyzed (Participants) | 98 | 57
  3 Months | 5.5 [0 to 51.5] | 12 [0 to 49]
  6 Months: number analyzed (Participants) | 98 | 52
  6 Months | 5 [0 to 60] | 21.5 [0 to 54.5]
  10 Months | 0 [0 to 8] | 0 [0 to 15]

11. Secondary Outcome: Treatment Engagement: Treatment Attendance Calendar (TAC)
Description: The TAC will be used to assess the total number of days treated for a substance abuse/mental health problem in the VA or other outpatient setting, 12-step or self-help group meetings, physician contacts and,hospitalization by treatment group. The TAC measure represent the total number of days experiencing any of these events by treatment group.
Time Frame: Weekly, 8 Weeks, 3 Months, 6 Months, 10 Months
Population: data are reported as those available at study baseline and each subsequent study outcome time point.
Measure: Median (Inter-Quartile Range); unit: days reported
Arm/Group | Mindfulness Based Relapse Prevention (MBRP): | Twelve-Step Facilitation Intervention (TSF)
Number analyzed (Participants) | 98 | 106
days reported
  Week 1: number analyzed (Participants) | 73 | 93
  Week 1 | 6 [0 to 13] | 4 [1 to 9]
  Week 2: number analyzed (Participants) | 69 | 78
  Week 2 | 4 [1 to 7] | 4 [1 to 6]
  Week 3: number analyzed (Participants) | 59 | 77
  Week 3 | 3 [1 to 7] | 3 [1 to 7]
  Week 4: number analyzed (Participants) | 51 | 68
  Week 4 | 3 [0 to 8] | 3 [2 to 6]
  Week 5: number analyzed (Participants) | 55 | 66
  Week 5 | 4 [1 to 7] | 4 [2 to 7]
  Week 6: number analyzed (Participants) | 50 | 62
  Week 6 | 4 [1 to 6] | 3 [1 to 6]
  Week 7: number analyzed (Participants) | 41 | 61
  Week 7 | 3 [1 to 4] | 3 [1 to 6]
  Week 8: number analyzed (Participants) | 52 | 68
  Week 8 | 3 [0 to 6] | 3 [1 to 6.5]
  3 Months: number analyzed (Participants) | 52 | 57
  3 Months | 8.5 [1.5 to 42] | 16 [3 to 45]
  6 Months: number analyzed (Participants) | 49 | 52
  6 Months | 4 [0 to 26] | 12 [2 to 34.5]
  10 Months: number analyzed (Participants) | 97 | 106
  10 Months | 0 [0 to 8] | 0 [0 to 10]

12. Secondary Outcome: Quality of Life Scale (QOLS) is a 16 Item Scale Measuring Quality of Life.
Description: This 16-item scale, used to assess satisfaction with major areas of life function, has convergent and discriminant construct validity in chronic illness as evidenced by high correlations between the QOLS total score and Life Satisfaction Index. Scores range from 1 = 112 with higher scores indicating higher satisfaction with quality of life.
Time Frame: Baseline, 8 Weeks, 3 Months, 6 Months, 10 Months
Population: Total Quality of life data from available measures at study treatment conclusion and at study follow up visits.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindfulness Based Relapse Prevention (MBRP): | Twelve-Step Facilitation Intervention (TSF)
Number analyzed (Participants) | 98 | 106
units on a scale
  Baseline: number analyzed (Participants) | 97 | 105
  Baseline | 74 (16) | 73 (18)
  Week 8: number analyzed (Participants) | 49 | 66
  Week 8 | 75 (16) | 81 (17)
  3 Months: number analyzed (Participants) | 51 | 56
  3 Months | 75 (15) | 80 (19)
  6 Months: number analyzed (Participants) | 49 | 52
  6 Months | 74 (17) | 80 (16)
  10 Months: number analyzed (Participants) | 52 | 53
  10 Months | 78 (16) | 80 (15)

13. Secondary Outcome: Urine Drug Screen - End of Study
Description: as for outcome 7
Time Frame: End of Study (up to 1 year)
Population: End of Study UDS results
Measure: Count of Participants; unit: Participants
Arm/Group | Mindfulness Based Relapse Prevention (MBRP): | Twelve-Step Facilitation Intervention (TSF)
Number analyzed (Participants) | 98 | 106
Participants
  THC: number analyzed (Participants) | 44 | 49
  THC | 8 | 6
  Coc: number analyzed (Participants) | 44 | 49
  Coc | 10 | 7
  PCP: number analyzed (Participants) | 44 | 49
  PCP | 0 | 1
  OPI: number analyzed (Participants) | 44 | 49
  OPI | 0 | 1
  MET: number analyzed (Participants) | 44 | 49
  MET | 1 | 0
  MTD: number analyzed (Participants) | 44 | 49
  MTD | 1 | 0
  AMP: number analyzed (Participants) | 44 | 49
  AMP | 1 | 0
  BAR: number analyzed (Participants) | 44 | 49
  BAR | 1 | 0
  BZO: number analyzed (Participants) | 44 | 49
  BZO | 0 | 1
  OXY: number analyzed (Participants) | 44 | 49
  OXY | 2 | 0
  MDMA: number analyzed (Participants) | 44 | 49
  MDMA | 0 | 0

14. Other Pre Specified Outcome: MINI-International Neuropsychiatric Interview
Description: The MINI is a well-standardized structured interview which is similar in sensitivity, specificity, and inter-rater reliability to other more lengthy diagnostic interviews, such as the Structured Clinical Interview for DSM-IV. A DSM-V version of the MINI is not available, so DSM-IV criteria will be utilized. The MINI will be used at baseline to assess psychiatric diagnoses for inclusion/exclusion and urn randomization purposes.
Time Frame: Baseline
Population: Baseline measure - all randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Mindfulness Based Relapse Prevention (MBRP): | Twelve-Step Facilitation Intervention (TSF)
Number analyzed (Participants) | 98 | 106
Participants
  MDE (Current) | 16 | 10
  MDE (Past) | 49 | 51
  MDD (Current) | 9 | 6
  MDD (Past) | 37 | 35
  Manic Episode (Current) | 4 | 3
  Manic Episode (Past) | 7 | 10
  Hypomanic Episode (Current) | 0 | 0
  Hypomanic Episode (Past) | 0 | 3
  Bipolar 1 (Current) | 0 | 0
  Bipolar 1 (Past) | 4 | 7
  Bipolar Unspec (Current) | 0 | 0
  Bipolar Unspec (Past) | 0 | 0
  Bipolar Unspec w/ Psych (Current) | 0 | 0
  Bipolar Unspec w/ Psych (Past) | 0 | 1
  Psychotic Disorder (Past Month) | 1 | 1
  Psychotic Disorder (Lifetime) | 1 | 7
  Mood Disorder w/ Psych (Current) | 1 | 1
  Mood Disorder w/ Psych (Lifetime) | 6 | 5
  Panic Disorder (Past Month) | 6 | 13
  Panic Disorder (Lifetime) | 10 | 18
  Agoraphobia (Current) | 16 | 11
  Social Anxiety (Current) | 16 | 12
  OCD (Current) | 4 | 3
  PTSD (Current) | 25 | 23
  AUD (Past 12 Mo) | 63 | 79
  SUD (Past 12 Mo) | 67 | 74

15. Other Pre Specified Outcome: Montreal Cognitive Assessment (MOCA)
Description: This brief, well-validated instrument will be used at baseline to screen for cognitive impairment that could interfere with ability to benefit from MBRP. A cut-off of 26/30 is considered normal. Scores range from 0 - 30 with lower scores indicating mores severe cognitive impairment.
Time Frame: Baseline
Population: Baseline Measure - all randomized participants
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindfulness Based Relapse Prevention (MBRP): | Twelve-Step Facilitation Intervention (TSF)
Number analyzed (Participants) | 98 | 106
units on a scale | 25.8 (2.6) | 25.9 (2.9)

16. Post Hoc Outcome: Study Visit Attendance
Description: Weekly study visit and follow-up visit attendance
Time Frame: Weekly, 8 Weeks, 3 Months, 6 Months, 10 Months
Population: all randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Mindfulness Based Relapse Prevention (MBRP): | Twelve-Step Facilitation Intervention (TSF)
Number analyzed (Participants) | 98 | 106
Participants
  Week 1 | 69 | 93
  Week 2 | 68 | 77
  Week 3 | 59 | 76
  Week 4 | 51 | 68
  Week 5 | 55 | 65
  Week 6 | 49 | 61
  Week 7 | 39 | 61
  Week 8 | 51 | 67
  3 Months | 50 | 55
  6 Months | 46 | 50
  10 Months | 47 | 50

ADVERSE EVENTS:
Time Frame: Study treatment, 8 weeks, follow-up, up to 10 months
Description: Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research. Adverse events were collected by self report assessment at baseline, weekly over the 8 week intervention, end of treatment and 3-, 6- and 10 months follow-up periods.
Arm/Group | Mindfulness Based Relapse Prevention (MBRP): | Twelve-Step Facilitation Intervention (TSF)
All-Cause Mortality (participants affected / at risk) | 1/98 | 1/106
Serious Adverse Events (participants affected / at risk) | 14/98 | 15/106
Other Adverse Events (participants affected / at risk) | 14/98 | 18/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Mindfulness Based Relapse Prevention (MBRP): (N=98) | Twelve-Step Facilitation Intervention (TSF) (N=106)
Relapse to Substance Use Disorder (Psychiatric disorders) | 7 (7) | 4 (4)
Depression (Psychiatric disorders) | 2 (4) | 4 (4)
Gallbladder surgery (Surgical and medical procedures) | 2 (2) | 0 (0)
Hernia surgery (Surgical and medical procedures) | 0 | 1/1
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chest Pain (Cardiac disorders) | 1 (1) | 0 (0)
iron defficiency (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Congestive Heart Failure (Cardiac disorders) | 0 (0) | 1 (1)
Occipital Fracture (Eye disorders) | 0 (0) | 1 (1)
Aneursym (Vascular disorders) | 1 (1) | 0 (0)
Homicidal Ideation (Psychiatric disorders) | 0 (0) | 1 (1)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
psychosis (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mindfulness Based Relapse Prevention (MBRP): (N=98) | Twelve-Step Facilitation Intervention (TSF) (N=106)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 5 (5)
urinary tract infection (Infections and infestations) | 1 (1) | 5 (5)
upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 6 (6)
Depression (Psychiatric disorders) | 4 (4) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-09-26): https://cdn.clinicaltrials.gov/large-docs/63/NCT02326363/Prot_SAP_000.pdf
  • Informed Consent Form (2016-06-01): https://cdn.clinicaltrials.gov/large-docs/63/NCT02326363/ICF_001.pdf